CLINICAL TRIAL: NCT05302843
Title: A Phase 1，Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Ascendind Doses of BPI-28592 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study of BPI-28592 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661211
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Metastasis, Neoplasm
Keywords: NTRK1/2/3, fusion
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose exploration and dose expansion (Experimental): Patients receive BPI-28592 PO. Cycles repeat every 28 days.
  Interventions: Drug: BPI-28592

INTERVENTIONS:
Drug: BPI-28592 — Characterize the pharmacokinetics (PK)，safety，antitumor activity of BPI-28592

SUMMARY:
This is an open-labe Phase I study of BPI-28592 for the treatment of patients with solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of locally advanced or metastatic solid tumor
* At least 18 years of age
* Measurable or evaluable disease
* Adequate organ function as defined per protocol

Exclusion Criteria:

* Symptomatic or unstable brain metastases
* Pregnancy or lactation
* Other protocol specified criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety and tolerability of BPI-28592 in subjects with advanced solid tumor malignancies | about 20 months
  Number of subjects with treatment related adverse events
determine the recommended Phase II dose (RP2D) and preliminarily to develop a suitable dosing regimen | about 20 months
  Number of subjects with dose limiting toxicity

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of BPI-28592 | about 20 months
  Blood plasma concentration
To determine overall response rate (ORR),calculated as the proportion of subjects with confirmed complete (CR) or partial response (PR) to BPI-28592 | about 20 months
  Evaluate clinical activity/efficacy of BPI-28592
To evaluate the duration of response (DOR) in subjects with CR or PR as best response | about 20 months
  Evaluate clinical activity/efficacy of BPI-28592
to evaluate the disease control rate (DCR) | about 20 months
  Evaluate clinical activity/efficacy of BPI-28592
To evaluate progression-free survival (PFS) following initiation of BPI-28592 | about 20 months
  Evaluate clinical activity/efficacy of BPI-28592
To evaluate overall (OS) following initiation of BPI-28592 | about 20 months
  Evaluate clinical activity/efficacy of BPI-28592

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Sheng J, Chen H, Fu B, Pan H, Wang J, Han W. BPI-28592 as a novel second generation inhibitor for NTRK fusion tumors. NPJ Precis Oncol. 2024 Sep 11;8(1):198. doi: 10.1038/s41698-024-00686-8. PMID 39256512